CLINICAL TRIAL: NCT01779076
Title: Emergence From General Anesthesia With Laryngeal Mask Airway and Increased End-expiratory Pressure Using 30% Oxygen is as Safe as With 100% Oxygen But Reduces the Area of Post Operative Atelectasis.
Brief Title: Oxygen Level and Safe Emergence From Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Lennart Edmark, M.D., Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr 2012 / 539
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Focus of Study is Postoperative Pulmonary Atelectacis
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100% oxygen during extubation (Experimental): In this arm the intervention will consist of 100 % oxygen.
  Interventions: Procedure: 100% oxygen
- 30% oxygen during extubation (Experimental): In this arm the intervention will consist of 30 % oxygen.
  Interventions: Procedure: 30% oxygen

INTERVENTIONS:
Procedure: 30% oxygen
  Arms: 30% oxygen during extubation
Procedure: 100% oxygen
  Arms: 100% oxygen during extubation

SUMMARY:
Using a protective ventilation strategy during general anesthesia from pre-oxygenation to emergence and selecting patients without risk of a difficult airway or intubation, a lower fraction of inspiratory oxygen (FIO2) can be used during extubation. This might reduce the postoperative area of atelectasis without desaturations becoming more common.

ELIGIBILITY:
Inclusion Criteria:

* No sign of difficult airway or intubation
* Day case surgery in total intravenous anesthesia with laryngeal mask airway without adding regional anesthesia of plexus brachialis or muscle relaxant.
* Body mass index less than 35.
* American Society of Anesthesiologists physical status (ASA) class I-III

Exclusion Criteria:

* Body mass index 35 or higher
* Increased risk of aspiration
* Obstructive sleep apnea syndrome
* Procedures during surgery making a former easy airway a difficult airway
* Need for opioids after extubation
* Hypothermia

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06-11 (Actual)

PRIMARY OUTCOMES:
Area of atelectasis | 30 minutes
  The area of atelectasis is investigated by computed tomography of the lungs postoperatively

SECONDARY OUTCOMES:
Peripheral oxygen saturation (SpO2) | 3 hours
  SpO2 is continuously assessed postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Enlund, M.D., Ph.D., Principal Investigator — Landstinget i Värmland
Locations (1):
- Västmanlands sjukhus Köping, Köping, Västmanland County, Sweden

REFERENCES:
- [Derived] Edmark L, Auner U, Lindback J, Enlund M, Hedenstierna G. Post-operative atelectasis - a randomised trial investigating a ventilatory strategy and low oxygen fraction during recovery. Acta Anaesthesiol Scand. 2014 Jul;58(6):681-8. doi: 10.1111/aas.12322. Epub 2014 Apr 11. PMID 24720763